CLINICAL TRIAL: NCT06714162
Title: A 12-week Randomized Controlled Clinical Trial Evaluating the Efficacy of a Dietary Supplement in an Adult Population.
Brief Title: A Dietary Supplement Examined for Anti-ageing Effects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prenetics Global (Industry)
Collaborators: San Francisco Research Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR20240502
Record Dates: First submitted 2024-11-04; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Ageing Signs
MeSH Terms: interventions — Longevity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): dietary supplement
  Interventions: Dietary Supplement: Longevity pill

INTERVENTIONS:
Dietary Supplement: Longevity pill — vitamins and herbs

SUMMARY:
dietary supplement for healthy ageing

ELIGIBILITY:
Inclusion Criteria: Healthy Adults -

Exclusion Criteria: Diseases deemed to be unable to participate in the study

-

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-21 (Estimated); Primary Completion 2025-02-27 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Cogntiion | 12 weeks
  Memory Test - Mini Mental State Exam where a higher score indicates a better memory

IPD SHARING:
Plan to Share IPD: Yes
de identified data excel spreadheets
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 11/21/2024 - 4/15/2025
Access Criteria: data excel sheets de identified through encrypted email